CLINICAL TRIAL: NCT07198802
Title: Molecular Research on Predictive Efficacy and New Therapeutic Targets for Nasopharyngeal Carcinoma Based on Tumor Immune Microenvironment
Brief Title: Molecular Research on Predictive Efficacy and New Therapeutic Targets for Nasopharyngeal Carcinoma
Status: Not yet recruiting | Type: Observational
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: WuhanUH 1149-01
Record Dates: First submitted 2025-07-17; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Nasopharyngeal Carcinoma (NPC)
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Study Groups
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This project involves no therapeutic intervention for the subjects.

SUMMARY:
To analyze the spatiotemporal dynamic evolution of nasopharyngeal carcinoma before and after immunotherapy and during tumor progression, 2~3 key cell subsets or node molecules were screened to predict the curative effect. Spatial metabolome and organoids were used to elucidate the mechanism of key factors leading to immunotherapy tolerance in NPC and identify new targets for intervention.

ELIGIBILITY:
Inclusion Criteria Before the trial, the participants must meet all of the following requirements to be eligible for inclusion.

1. Clearly diagnosed with nasopharyngeal carcinoma by pathology;
2. Patients who have received combined radiotherapy, chemotherapy and immunotherapy in our hospital;
3. Patients diagnosed in our hospital from January 2025 to December 2028;
4. Have relatively complete clinical data;
5. Age between 15 and 75 years old;

Exclusion Criteria Before the trial, the participants who meet any of the following requirements cannot be included.

1. The final diagnosis of the participants is other diseases, including lymphoma, or oropharyngeal cancer, etc.;
2. The participants failed to obtain pathological and imaging data for various reasons;
3. Due to physical conditions, they did not undergo relevant examinations, refused to accept examinations, or interrupted treatment for other reasons, and were unable to complete clinical assessment.

Ages: 15 Years to 75 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with nasopharyngeal carcinoma who were admitted to our hospital
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Failure-free survival (FFS) | 3-year
  Failure-free survival is measured from day of diagnosis until treatment failure, death from any cause, or last follow-up visit, whichever occurred first

SECONDARY OUTCOMES:
Overall survival (OS) | 5-year
  Overall survival is measured from day of diagnosis until death due to any cause or the latest known date alive